CLINICAL TRIAL: NCT06142669
Title: Post Market Clinical Follow-Up Study for EVOLUTION® Revision Tibial System and EVOLUTION® Stemmed CS Femur With the EVOLUTION® MP CS Tibial Insert
Brief Title: EVOLUTION® Revision STEMMED CS Post Market Clinical Follow-up Study Protocol
Status: Recruiting | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18K001CS
Record Dates: First submitted 2023-05-24; First posted 2023-11-21 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-11

CONDITIONS: Joint Diseases
Keywords: Knee Osteoarthritis; Revision Procedure; Knee arthroplasty
MeSH Terms: conditions — Joint Diseases; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Revision Total Knee Arthroplasty: Single study group with either newly or previously implanted subjects with the EVOLUTION® Revision Tibia and EVOLUTION® Revision STEMMED CS Femur with the EVOLUTION® MP CS Insert.
  Interventions: Device: EVOLUTION® Revision Tibial System and EVOLUTION® Stemmed CS Femur with the EVOLUTION® MP CS Tibial Insert

INTERVENTIONS:
Device: EVOLUTION® Revision Tibial System and EVOLUTION® Stemmed CS Femur with the EVOLUTION® MP CS Tibial Insert — Primary knee arthroplasty or a revision knee that requires a revision procedure.

SUMMARY:
MicroPort (MPO) is conducting this PMCF study to evaluate the safety and effectiveness of its EVOLUTION® Revision Tibial System and EVOLUTION® Revision STEMMED CS Femur with the EVOLUTION® MP CS Tibial Insert. This type of study is required by regulatory authorities for all devices that have been approved in Europe to evaluate the medium and long-term clinical evidence.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate individual component survivorship for tibial base, femoral component, and tibial insert at specified intervals out to 10 years follow-up.

The secondary objectives include:

* Determine the cumulative incidence of individual component revision at specified intervals out to 10 years follow-up;
* Characterize functional scores for subjects, as assessed by KOOS Scores and EQ-5D-5L Scores, out to 10 years follow-up;
* To assess subject satisfaction with their TKA procedure using the Forgotten Joint Score and a Satisfaction Survey;
* To assess the presence, zone, and the size of radiolucencies surrounding implanted components out to 10 years follow-up;
* To assess safety and characterize protocol defined adverse events and adverse device effects.

ELIGIBILITY:
Inclusion Criteria:

1. Has previously undergone or currently has been determined to undergo a revision knee arthroplasty that requires implantation of the components under study (EVOLUTION® Revision Tibial System and EVOLUTION® STEMMED CS Femur with the EVOLUTION® MP CS Tibial Insert)
2. Decision to perform the study index surgery with the required study components is pre-determined regardless of the research;
3. Previously implanted subjects must be enrolled within 3 years (+ 6 months) of their study index surgery
4. Willing to voluntarily sign the informed consent form
5. Willing and able to comply with the protocol, able to read and complete the required forms, and willing and able to adhere to the requirements of the protocol through the 10-year postoperative follow-up visit.

Exclusion Criteria:

1. Skeletally immature (less than 21 years of age) at time of implantation
2. Has or had an overt infection at the time of implantation
3. Has or had inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable
4. Currently enrolled in another clinical investigation which could affect the endpoints of this protocol
5. Has or had documented substance abuse issues
6. Has or had an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
7. Currently incarcerated or has impending incarceration
8. Has a medical condition, as judged by the Investigator, that would interfere with the subject's ability to comply with the requirements of the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter, prospective follow-up study of newly or previously implanted subjects. Previously implanted subjects must be enrolled within 3 years (+ 6 months) of the study index surgery.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2036-06 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of EVOLUTION® Revision Tibial Base components survivorship out to 10 years. | up to 10 years
  Percentage of knees survived with no revision or replacement at 10-year
The proportion of EVOLUTION® STEMMED CS Femoral components survivorship out to 10 years. | up to 10 years
  Percentage of knees survived with no revision or replacement at 10-year
The proportion of EVOLUTION® MP CS tibial inserts survivorship out to 10 years. | up to 10 years
  Percentage of knees survived with no revision or replacement at 10-year

SECONDARY OUTCOMES:
Functional Scores | Year 1,Year 3, Year 5, Year 7, and Year 10
  To assess functional scores utilizing Knee Injury and Osteoarthritis Outcome Score (KOOS Scores) out to 10 years follow-up.
Functional Scores | Year 1,Year 3, Year 5, Year 7, and Year 10
  To assess subject satisfaction with their Total Knee Arthroplasty (TKA) procedure utilizing the Forgotten Joint Score (FJS) at specified intervals out to 10 years follow-up.
Functional Scores | Year 1,Year 3, Year 5, Year 7, and Year 10
  To assess functional scores utilizing EQ-5D-5L at specified intervals out to 10 years follow-up.
Subject Satisfaction | Year 1,Year 3, Year 5, Year 7, and Year 10
  To assess subject satisfaction with their TKA procedure via the Satisfaction Survey at specified intervals out to 10 years follow-up.
Radiolucencies | Year 1,Year 3, Year 5, Year 7, and Year 10
  To assess the presence of radiolucencies surrounding the implanted components at specified intervals out to 10 years follow-up.
To assess subject safety: Adverse Events o Adverse Events related to study device or the index surgical procedure | Year 1,Year 3, Year 5, Year 7, and Year 10
  To assess safety and characterize protocol defined adverse events and adverse device effects.
Incidence of component revision | Year 1,Year 3, Year 5, Year 7, and Year 10
  Determine the cumulative incidence of individual component revision at specified intervals out to 10 years follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pietro I Randelli, Prof, Principal Investigator — Gaetano Pini Orthopedic Institute
Locations (1):
- Gaetano Pini Orthopedic Institute, Milan, Piazza C. Ferrari 1 20122 Milan, Italy